CLINICAL TRIAL: NCT01679015
Title: Concomitant Dry Eye in Patients With Ocular Allergy: an Under Recognized and Poorly Managed Syndrome
Brief Title: Evaluating Patients With Eye Allergies and Determining if There Are Also Dry Eyes
Status: Completed | Type: Observational
Sponsor: Schwartz Laser Eye Center (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Marc R.Bloomenstein, O.D., Schwartz Laser Eye Center
Other Study IDs: AL-001
Record Dates: First submitted 2012-08-20; First posted 2012-09-05 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2013-01

CONDITIONS: Dry Eyes; Allergic Conjunctivitis
Keywords: Burning; Dryness; Itching; Blurry Vision
MeSH Terms: conditions — Dry Eye Syndromes; Conjunctivitis, Allergic; Paresthesia; Pruritus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dry Eyes, Eye Allergies: Patients with ocular allergies and those with dry eyes.

SUMMARY:
Evaluating the percentage of patients that suffer from eye allergies and determining whether they also have dry eyes.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Males and females at least 18 years of age
* Personal history of allergic disorders including but not limited to allergic conjunctivitis, allergic rhinitis, contact dermatitis and other eczema, and asthma
* Diagnosis of allergic conjunctivitis
* Presence of any of the following signs including conjunctival redness and papillae, chemosis, red edematous eyelids, reduced tear clearance, reduced TBUT, vital staining, stringy discharge, and/or symptoms including ocular itching, burning and tearing, runny nose or itchy throat

Exclusion Criteria:

* Active ocular or systemic infection
* History of ocular infection within past 6 months
* Presence of punctal plugs
* Recent ocular surgery within past 6 months
* Current use of chemotherapeutic agents
* Presence of ocular trauma
* Inability to give informed consent
* Women who are pregnant, nursing or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be screened from existing patient database.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2012-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Prevalence of dry eye in an allergic population presenting to a high volume optometry practice | up to 2 years

SECONDARY OUTCOMES:
Prevalence of allergic patients with moderate to severe ocular signs and symptoms | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Marc R Bloomenstein, O.D., Principal Investigator — Schwartz Laser Eye Center
Locations (1):
- Schwartz Laser Eye Center, Scottsdale, Arizona, United States